CLINICAL TRIAL: NCT05812456
Title: Comparison of Shear Bond Strength of Different Commercial Brands of Stainless Steel Orthodontic Brackets: An in Vitro Study
Brief Title: Comparison Between Shear Bond Strength of Different Commercial Metal Bracket Brands: an in Vitro Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Mostafa Hamdy Mohamed Afifi, Principle investigator, Future University in Egypt
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FUE.REC(29)/12/2020
Record Dates: First submitted 2023-03-15; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Orthodontic Appliance Complication; Shear Strength
Keywords: Orthodontic brackets brands; Shear bond strength; Remanent adhesive Index

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: this is a double-blinded study (investigator-outcome assessor) this is a double-blinded study, for both the investigator and outcome assessor, as the investigator will be responsible for collecting the sample and preparing the sample for the experiment.
  The outcome assessors will be blinded during the intervention application. as he/she will be responsible for analyzing the results of each group in the experiment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 3m Metal Brackets (Active Comparator): 3m Unitek Gemini Roth Stainless-Steel Brackets. it is passive Stainless-Steel components used in fixed Orthodontics appliance to help in solving malocclusions by bonding it to teeth's enamel. it acts as a means to transfers forces applied by activated archwires inserted in bracket slots to try to correct and improve the patients malocclusion problems.
  There are different sizes of Stainless-Steel bracket slots, There are 0.018 slot and 0.022 slot.
  Brackets are made of many different materials such as Stainless-Steel, ceramics, plastic or 3d printed. The most used type is metal brackets.
  Brackets come with built in prescriptions of torque and tip, there are two type of prescriptions: Roth and MBT
  Interventions: Other: Estimation of Shear Bond Strength
- American Orthodontics Metal Brackets (Active Comparator): American Orthodontics Mini Masters 0.022 Roth Stainless-Steel Brackets. it is passive Stainless-Steel components used in fixed Orthodontics appliance to help in solving malocclusions by bonding it to teeth's enamel. it acts as a means to transfers forces applied by activated archwires inserted in bracket slots to try to correct and improve the patients malocclusion problems.
  There are different sizes of Stainless-Steel bracket slots, There are .18 slot and .22 slot.
  Brackets are made of many different materials such as Stainless-Steel, ceramics, plastic or 3d printed. The most used type is metal brackets.
  Brackets come with built in prescriptions of torque and tip, there are two type of prescriptions: Roth and MBT
  Interventions: Other: Estimation of Shear Bond Strength
- Fanta Metal Brackets (Experimental): Fanta Firmax 0.022 Roth Stainless-Steel Brackets. Fanta is a Chinese Orthodontic bracket brand that started to spread.
  it is passive Stainless-Steel components used in fixed Orthodontics appliance to help in solving malocclusions by bonding it to teeth's enamel. it acts as a means to transfers forces applied by activated archwires inserted in bracket slots to try to correct and improve the patients malocclusion problems.
  There are different sizes of Stainless-Steel bracket slots, There are 0.018 slot and 0.022 slot.
  Brackets are made of many different materials such as Stainless-Steel, ceramics, plastic or 3d printed. The most used type is metal brackets.
  Brackets come with built in prescriptions of torque and tip, there are two type of prescriptions: Roth and MBT
  Interventions: Other: Estimation of Shear Bond Strength
- Matt Orthodontics Metal Brackets (Experimental): Matt Orthodontics Pierre 0.022 Roth Metal Brackets. Matt is a Chinese Orthodontic bracket brand that started to spread.
  it is passive Stainless-Steel components used in fixed Orthodontics appliance to help in solving malocclusions by bonding it to teeth's enamel. it acts as a means to transfers forces applied by activated archwires inserted in bracket slots to try to correct and improve the patients malocclusion problems.
  There are different sizes of Stainless-Steel bracket slots, There are 0.018 slot and 0.022 slot.
  Brackets are made of many different materials such as Stainless-Steel, ceramics, plastic or 3d printed. The most used type is metal brackets.
  Brackets come with built in prescriptions of torque and tip, there are two type of prescriptions: Roth and MBT
  Interventions: Other: Estimation of Shear Bond Strength

INTERVENTIONS:
Other: Estimation of Shear Bond Strength — Measuring shear bond strength between the different bracket brands and the enamel will be estimated by aiming the edge of the blade of the universal testing machine at bracket-enamel interface. The force required to debond each bracket will be registered in Newtons (N), and converted to Megapascals by dividing the force registered in newtons on each bracket base area (mm2).
  After bond failure, the brackets and the enamel surfaces will be examined and assessed for the amount of adhesive remaining on the bracket bases by using digital microscope at 35x magnification. this will identify the site of bond failure.
  Other Names: Evaluation of Adhesive Remnant Index

SUMMARY:
some orthodontic brands are more expensive than others, one of the primary outcomes of this study is to know if is it worth using expensive brands? will it provide better quality treatment, in particular, bond strength? The treatment duration is long therefore it is expensive, either for the orthodontist and/or the patient.

This study will be comparing the bond strength of different commercial brands of stainless steel brackets.

DETAILED DESCRIPTION:
There are a plethora of studies in the science of orthodontics discussing different massive advances in the orthodontic adhesion concepts that allowed orthodontists to successfully bond brackets and tubes to teeth. the bond strength between the bracket and tooth should be sufficient to withstand the forces of mastication and the aggressive conditions of the oral environment. a commonly encountered problem is the failure of the bond between the bracket and tooth during treatment.

There are a lot of orthodontic in vitro studies that discussed bond failure and strength. multiple studies have studied the bracket-enamel bond strength with different curing systems and found that there was no significant difference in terms of bond strength. Several other studies discussed the effect of different adhesive systems on the bond strength to the enamel.

There are many studies that debated the shear bond strength of different metal bracket base shapes and sizes concluding that no differences in SBS for the surface area within the range of 6.82-12.35mm2 as well as the shape of the bracket base had no effect on shear bond strength.

The effectiveness or the success of the orthodontic treatment is arbitrated by achieving better aesthetics, better function, and better judgment for the patient too.

Even if there was a plethora of studies comparing the bond strength of different bracket shapes and sizes and also between metal and ceramic brackets, however, none have considered comparing shear bond strength of different bracket brands to enamel, Considering its cost and repeated failure which has its implication on both patient and orthodontist.

ELIGIBILITY:
Inclusion Criteria:

* sound extracted upper and/or lower permanent premolars.
* Intact buccal enamel surface with n erosion and cracks.
* the teeth must be free from caries, restoration, white spot lesions, or any sign of decalcification.
* No pretreatment with any chemical agents such as hydrogen peroxide or formalin.

Exclusion Criteria:

* teeth with amelogenesis or dentinogenesis imperfecta.
* labially restored teeth.
* endodontically treated teeth.
* teeth with fluorosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Estimation of Shear Bond Strength | 24 hours
  Measuring shear bond strength between the different bracket brands and the enamel will be estimated by aiming the edge of the blade of the universal testing machine at bracket-enamel interface. The force required to debond each bracket will be registered in Newtons (N), and converted to Megapascals by dividing the force registered in newtons on each bracket base area (mm2).

SECONDARY OUTCOMES:
Evaluation of Adhesive Remanent Index | 24 hours
  ARI scale is used to asses site of bond failure After bond failure, the brackets and the enamel surfaces will be examined and assessed for the amount of adhesive remaining on the bracket bases by using digital microscope at 35x magnification.

CONTACTS AND LOCATIONS:
Locations (1):
- Future Unversity in Egypt, New Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided